CLINICAL TRIAL: NCT04358159
Title: Randomised Controlled Trial of Ventralex Versus Onlay Mesh Repair for Midline Incisional Hernias
Brief Title: RCT Ventralex vs Onlay Mesh in Incisional Hernias
Acronym: VPatchIncRCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gabriel Sandblom, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VPatchIncRCT
Record Dates: First submitted 2020-04-19; First posted 2020-04-24 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Incisional Hernia of Midline of Abdomen

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial of Vantralex versus Progrip for repair of midline incisional hernias
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and staff responsible for the postoperative care of the patient are masked to the acollcation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ventralex (Experimental): Repair with Ventralex patch in sublay position
  Interventions: Device: Ventralex
- Progrip (Active Comparator): Repair with Progrip in Onlay position
  Interventions: Device: Progrip

INTERVENTIONS:
Device: Ventralex — Repair of the hernia by a Ventralex patch in sublay position
  Arms: Ventralex
Device: Progrip — Repair of the hernia by a Progrip mesh in onlay position
  Arms: Progrip

SUMMARY:
A radomised controlled trial comparing Ventralex patch and Progrip mesh in surgery for midline incisional hernias

DETAILED DESCRIPTION:
Incisional hernias in the midline is among the most common conditions requiring surgery. There are several factors which can increase the risk of incisional hernias, e.g. surgical technique, truncal obesity and other co-morbidities.

Repair with mesh-reinforcement is considered standard for the treatment of incisional hernias. Onlay and sublay mesh placements are the most commonly used methods. There are many different types of mesh available to use. Despite the widely use of composite ventral-patch Ventralex, there are few studies with small numbers of patients showing the advantage and disadvantage of ventral-patch. Some studies show that the onlay mesh-reinforcement remains a good alternative to the sublay mesh technique, while others showing fewer recurrences with the sublay mesh technique. The Ventralex mesh is usually placed on the peritoneum as a Intra peritoneum onlay mesh (IPOM). In this study intend to compare pre peritoneal Ventralex® mesh in sublay position with ProGrip self-fixating onlay mesh.

ELIGIBILITY:
Inclusion Criteria:

* Hernia defect 1-4 cm
* Incisional hernia or recurrent hernia after previous primary hernia repair
* BMI <35
* Age 18-100 years

Exclusion Criteria:

* Defect size>4 cm
* Ongoing pregnancy
* BMI>35
* Primary hernia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | One year
  Rate of hernia recurrences diagnosed at clinical and/or radiologic examination

SECONDARY OUTCOMES:
Rate ofntra- and postoperative complications | 30 days
  Rate of complications occurring during or after the repair
Rate of seroma | one year
  Postoperative seroma
Persisting postoperative pain | One year
  Pain interfering with daily activities as rated with Ventral Hernia Pain Questionnaire
Sick leave | 30 days
  Mean number of postoperative days sick leave

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Sandblom, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karlskoga Hospital, Karlskoga, Sweden

IPD SHARING:
Plan to Share IPD: No